CLINICAL TRIAL: NCT02435927
Title: Phase I Study to Evaluate the Safety and Tolerability of ASLAN001 in Combination With Oxaliplatin and Capecitabine or Oxaliplatin and 5-FU With Leucovorin
Brief Title: ASLAN001 in Combination With Oxaliplatin and Capecitabine or Oxaliplatin and 5-FU With Leucovorin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: ASLAN Pharmaceuticals (Other); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-002SG
Record Dates: First submitted 2015-04-23; First posted 2015-05-06 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASLAN001 + CAPOX (Experimental): ASLAN001 + CAPOX: ASLAN001 twice daily in combination with oxaliplatin 130 mg/m2 intravenously on day 1 and capecitabine 850 mg/m2 orally twice daily on days 1 to 14 every 3 weeks
  Interventions: Drug: ASLAN001+ CAPOX (Oxaliplatin, capecitabine)
- ASLAN001 + mFolfox6 (Experimental): ASLAN001 + mFolfox6: ASLAN001 twice daily in combination with mFolfox6 (oxaliplatin 85 mg/m2 intravenously on day 1 and 5-FU bolus 400mg/m2 i.v on day 1 and as a continuous infusion 2400mg/ m2 over 46h and leucovorin 400mg/2 i.v on day 1) every 2 weeks
  Interventions: Drug: ASLAN001 + mFolfox6 (5-FU, leucovorin)

INTERVENTIONS:
Drug: ASLAN001+ CAPOX (Oxaliplatin, capecitabine) — ASLAN001 in combination with oxaliplatin and capecitabine
  Other Names: eloxatin, xeloda
  Arms: ASLAN001 + CAPOX
Drug: ASLAN001 + mFolfox6 (5-FU, leucovorin) — ASLAN001 in combination with 5-FU and leucovorin
  Other Names: 5-Fluorouracil, Folinic acid
  Arms: ASLAN001 + mFolfox6

SUMMARY:
This is a Phase I, open-label, dose escalation study of ASLAN001 given in combination with CAPOX or mFolfox6, in patients with metastatic solid tumours, whom are suitable to receive CAPOX or mFolfox6, or with tumours that have dysregulated EGFR or HER2 signaling.

DETAILED DESCRIPTION:
The study will use standard 3+3 design to determine the MTD (maximum tolerated dose) of ASLAN001 in combination with fixed dose of Oxaliplatin/Capecitabine (CAPOX) or 5-FU/leucovorin (mFolfox6).

MTD of ASLAN001 in combination with CAPOX will first be determined followed by the combination with mFolfox6.

The recommended Phase II dose will be the highest dose of the combination therapy that is considered to be tolerated in 6 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic solid tumours eligible for treatment with oxaliplatin in combination with capecitabine / 5-FU (fluorouracil) and leucovorin or who progressed following standard therapy or patients with EGFR (epidermal growth factor receptor ) or HER2 dysregulated tumours.
2. Patients with a partial gastrectomy may be allowed to participate in the study as long as they can take oral medications and meet all other inclusion/exclusion criteria.
3. Eastern Cooperative Oncology Group performance status of 0 or 1.
4. Adequate organ and hematological function as evidenced by the following laboratory studies within 14 days prior to enrolment:

   • Hematological function, as follows: Absolute neutrophil count ≥ 1.5 x 109/L. Platelet count ≥ 100 x 109/L. Hemoglobin ≥ 9 g/dL.

   • Coagulation function, as follows: Prothrombin time and activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN) per institutional laboratory normal range.

   • Renal function, as follows: Creatinine clearance ≥ 50 mL/min as calculated by Cockcroft-Gault formula.

   • Hepatic function, as follows: Total bilirubin ≤ 1.5 x ULN. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present).
5. Patients undergoing mandatory biopsy in dose expansion of a non-DLT cohort should have any of the following:

   * known HER2 or EGFR dysregulation
   * Patients with T790M mutation will be excluded.
   * Co-expression of HER2 and EGFR
6. Archival tumour sample is available for molecular profiling, unless undergoing tumour biopsy as part of the trial.

Exclusion Criteria:

1. Patients with persistent gastric outlet obstruction, complete dysphagia or feeding jejunostomy.
2. Patients receiving proton pump inhibitors or H2 antagonists for established, symptomatic gastro duodenal ulceration or gastroesophageal reflux disease. H2 antagonist can be prescribed after DLT (dose-limiting toxicity) period (the first 2 cycles) at the discretion of the investigator.
3. Patients with unresolved toxicities of grade 2 or more from prior anti-cancer therapies excluding alopecia.
4. Untreated or symptomatic central nervous system metastases. Patients with treated brain metastases stable for 3 months are eligible to enroll.
5. Major surgical procedures within 28 days prior to enrolment.
6. Clinically significant cardiovascular diseases that are symptomatic or uncontrolled.
7. Known active infection for human immunodeficiency virus, hepatitis B and C.
8. Pregnant or breast-feeding females.
9. Treatment with any of the following anti-cancer therapies prior to the first dose of study drugs within the stated timeframes

   * Cyclical chemotherapy within a period of time that is shorter than the cycle length used for that treatment. Exception for weekly chemotherapy regimens, where a minimum of 2 week washout from the last dose is required.
   * Biological therapy (e.g., antibodies) within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks, whichever is shorter, prior to starting study drug
   * Continuous or intermittent small molecule therapeutics within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug
   * Any other investigational agents within a period of time that is ≤ 5 t1/2 or less than the cycle length used for that treatment or ≤ 4 weeks (whichever is shortest) prior to starting study drug
   * Wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug
   * Previous combination therapy with xeloda and oxaliplatin within 6 months of study treatment.
   * Previous combination therapy with Oxaliplatin, 5-FU and Leucovorin (mFolfox6) within 6 months of study treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ASLAN001 when used in combination with Oxaliplatin and Capecitabine (CAPOX) or Oxaliplatin and 5-FU with leucovorin (mFolfox6) | one year

SECONDARY OUTCOMES:
Pharmacokinetic parameter Area under the plasma concentration time curve (AUC) | Day 1 and Day 15 of Cycle 1 and Day 1 of Cycle 3
Pharmacokinetic parameter Maximum plasma concentration (Cmax) | Day 1 and Day 15 of Cycle 1 and Day 1 of Cycle 3
Pharmacokinetic parameter Minimum (trough) plasma concentration (Cmin) | Day 1 and Day 15 of Cycle 1 and Day 1 of Cycle 3
Efficacy of ASLAN001 when given in combination in CAPOX or mFolfox6 as measured by the objective response rate (ORR) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew CH Ng, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore